CLINICAL TRIAL: NCT07346456
Title: Intraocular Lens Power Calculation Formulas in Eyes With Posterior Corneal Elevation ≥15 µm: An Eyetemis-based Comparative Analysis
Brief Title: Comparison of IOL Formulas in Eyes With PCE≥15µm
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Shen Weichen, Ophthalmology resident, Second Affiliated Hospital of Xi'an Jiaotong University
Other Study IDs: 3123315445
Record Dates: First submitted 2026-01-02; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-09

CONDITIONS: The Comparison of IOL Formulas in Eyes With PCE≥15um Undergoing Cataract Surgery
Keywords: IOL formulas; posterior corneal elevation; refractive outcomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intraocular lens calculation formulas — The study evaluates four groups of intraocular lens (IOL) power calculation formulas, totaling 13 distinct formulas, to compare their accuracy in predicting postoperative refractive outcomes in cataract patients.
  Group 1 - Without PK: Barrett Universal II (BUⅡ), EVO 2.0, Kane, Hill-RBF 3.0, LADAS, Pearl-DGS, and K6, which do not incorporate PK.
  Group 2 - Measured PK-I: Barrett TK measured (I) and EVO Advanced (I), which use measured PK from IOLMaster 700.
  Group 3 - Measured PK-P: Barrett TK measured (P) and EVO Advanced (P), which use measured PK from Pentacam AXL.
  Group 4 - Predicted PK: Barrett TK predicted and Kane KC, which estimate PK through prediction algorithms rather than direct measurement.
  This observational study does not introduce experimental procedures; all data are collected during routine cataract surgery and postoperative follow-up to determine the comparative accuracy of these formulas

SUMMARY:
The goal of this observational study is to evaluate the long-term refractive outcomes of advanced intraocular lens (IOL) power calculation formulas in cataract patients with posterior corneal elevation (PCE ≥ 15 μm).

The main question it aims to answer is:

Do PK-based formulas provide superior refractive accuracy compared with Without-PK-based formulas in patients with elevated posterior corneal surfaces?

Participants undergoing routine cataract surgery will have their biometry measured by both Pentacam AXL and IOLMaster 700, and postoperative refraction will be collected at 1 month, 3 months, and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the indications for cataract surgery, and undergoing Phacoemulsification + IOL implantation performed by the same surgeon.
* Preoperative biometry performed with IOLMaster 700 and Pentacam AXL, with a posterior corneal elevation greater than 15 μm within the central 5 mm zone on Scheimpflug imaging, and a central corneal thickness > 500 μm.
* Surgery completed successfully without any intraoperative or postoperative complications.
* Postoperative subjective refraction performed at 1 month after surgery by the same experienced optometrist.

Exclusion Criteria:

* Patients with pterygium, corneal diseases, glaucoma, uveitis, or fundus diseases (such as macular edema, retinal detachment), excluding high myopia.
* History of ocular trauma or previous intraocular surgery.
* Occurrence of intraoperative or postoperative complications, such as iris injury, posterior capsule rupture, IOL dislocation, vitreous prolapse, or vitreous hemorrhage.
* Postoperative best corrected visual acuity (BCVA) worse than 0.5.
* Difference between postoperative subjective refraction and preoperative target refraction greater than 2.00 D.
* Incomplete measurement data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 2024 to January 2025, patients who visited our hospital, were diagnosed with age-related cataract, and underwent cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
absolute SEQ-PE(accuracy) | From enrollment to the end of treatment at 6 months
  the absolute values of SEQ-PE
SEQ-PE(trueness) | From enrollment to the end of treatment at 6 months
  Spherical Equivalent Prediction Error
  1. SEQ=Sphere+2Cylinder
  2. PE=Postoperative Manifest SEQ-Predicted SEQ
Precision | From enrollment to the end of treatment at 6 months
  Precision refers to the consistency of the prediction errors (PE) of a formula across a study population, indicating how closely the individual prediction errors cluster around the central tendency (e.g., mean or median). A formula with higher precision shows smaller variability in its prediction errors.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Bai, Study Director — Department of Ophthalmology, The Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Department of Ophthalmology, The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No